CLINICAL TRIAL: NCT03197233
Title: Norwegian Mother and Child Study - Causal Pathways for Asthma (CASPAR)
Brief Title: Vitamin A and D Intake in Pregnancy, Infant Supplementation and Asthma Development
Status: Completed | Type: Observational
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Other Study IDs: PDB532_journal 08/2602-29; 221097 (Other Grant/Funding Number: Norwegian Research Council/BIOBANK program); ZO1ES49019 (Other Grant/Funding Number: National Institute of Environmental Health Sciences)
Record Dates: First submitted 2017-06-19; First posted 2017-06-23 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Asthma in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Maternal vitamin A and D intake during pregnancy — Dietary exposures during pregnancy and infant supplement use were assessed from maternal questionnaire report
  Other Names: Total vitamin A and D intake from food and supplements

SUMMARY:
The objective of this study is to investigate if maternal intake of vitamins A and D from food and dietary supplements during pregnancy, and infant supplementation with these vitamins, are associated with development of asthma in the offspring.

DETAILED DESCRIPTION:
This study was conducted as part of the research project "Causal pathways for asthma" funded by the Norwegian Research Council (2013-2017). The overall objective was to study if different pregnancy and early life exposures affect the risk of asthma and allergic diseases in children, and if these exposures exert their effects through epigenetic mechanisms, more specifically DNA methylation.

For this project, including the current study, existing data from the Norwegian Mother and Child Study (MoBa file version 9, 115 398 children and 95 248 mothers) were linked with the Medical Birth Registry of Norway and the Norwegian Prescription Database. The MoBa study recruited pregnant women between 1999 and 2008, at approximately 18 weeks of gestation. Beginning 2002, women completed a food frequency questionnaire about dietary intake (food and supplements) in pregnancy. A panel of maternal plasma biomarkers, including plasma retinol and 25-hydroxyvitamin D2 and D3, was available for a random sample of around 3,000 women who gave birth in 2002 and 2003.

ELIGIBILITY:
Inclusion Criteria:

Available maternal dietary intake data from pregnancy. Child turned 7 years by July 1st 2014.

Exclusion Criteria:

No maternal baseline questionnaire. Maternal energy intake <4,500 or > 20,000 kJ. No dietary supplement data. No linkage to national birth registry, or non-live births, or multiple births. Child death, or emigration, or unknown vital status.

Ages: 7 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The Norwegian Mother and Child Study is a population-based pregnancy cohort (births 1999-2009). Women were recruited nationwide (41% participation) around 18 weeks gestation. The current study included 61,676 eligible chidren born 2002-2007.
Sampling Method: Non-Probability Sample
Enrollment: 61676 (Actual)
Dates: Start 1999-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Child asthma based on dispensed asthma medications | A minimum of two dispensations around age 7 years
  Dispensations of antiasthmatics (Anatomical Therapeutic Chemical Classification/ATC codes R03AC, R03BA, R03AK, and R03DC) registered in the Norwegian Prescription Database

CONTACTS AND LOCATIONS:
Overall Officials: Wenche Nystad, PhD, Principal Investigator — Dept of Non-Communicable Diseases, Norwegian Institute of Public Health

IPD SHARING:
Plan to Share IPD: Yes
Data have been shared with collaborators.

REFERENCES:
- [Background] Magnus P, Birke C, Vejrup K, Haugan A, Alsaker E, Daltveit AK, Handal M, Haugen M, Hoiseth G, Knudsen GP, Paltiel L, Schreuder P, Tambs K, Vold L, Stoltenberg C. Cohort Profile Update: The Norwegian Mother and Child Cohort Study (MoBa). Int J Epidemiol. 2016 Apr;45(2):382-8. doi: 10.1093/ije/dyw029. Epub 2016 Apr 10. PMID 27063603
- [Background] Ronningen KS, Paltiel L, Meltzer HM, Nordhagen R, Lie KK, Hovengen R, Haugen M, Nystad W, Magnus P, Hoppin JA. The biobank of the Norwegian Mother and Child Cohort Study: a resource for the next 100 years. Eur J Epidemiol. 2006;21(8):619-25. doi: 10.1007/s10654-006-9041-x. Epub 2006 Sep 20. PMID 17031521
- [Derived] Parr CL, Magnus MC, Karlstad O, Holvik K, Lund-Blix NA, Haugen M, Page CM, Nafstad P, Ueland PM, London SJ, Haberg SE, Nystad W. Vitamin A and D intake in pregnancy, infant supplementation, and asthma development: the Norwegian Mother and Child Cohort. Am J Clin Nutr. 2018 May 1;107(5):789-798. doi: 10.1093/ajcn/nqy016. PMID 29722838